CLINICAL TRIAL: NCT06459817
Title: Quantitative Assessment of BB-02 Therapy Effect on Cartilage Status in Patients Affected by Early Knee Osteoarthritis
Acronym: JOCARE-OA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JOCARE-OA
Record Dates: First submitted 2024-05-23; First posted 2024-06-14 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis, Knee
Keywords: knee; osteoarthritis; preserving treatment; mri; Biophysical stimulation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 (Experimental): BB-02 therapy. 1h a day for 3 months
  Interventions: Device: BB-02 therapy
- group 2 (Experimental): BB-02 therapy. 4h a day for 1 month
  Interventions: Device: BB-02 therapy

INTERVENTIONS:
Device: BB-02 therapy — Biophysical stimulation with magnetic fields

SUMMARY:
Knee osteoarthritis is a condition that affects young or middle-aged patients with high functional demands. Knee replacement surgery in patients under 65 years of age is associated with a high risk of failure and the need for revision. For this reason, it becomes crucial to identify treatment alternatives aimed primarily at resolving symptoms but also at slowing down the joint degenerative process, with the goal of delaying the need for prosthetic treatment as much as possible. The medical device BB-02 (IGEA SpA, Carpi, Italy) is a certified medical device according to Regulation (EU) 2017/745 (MDR) for the treatment of inflammatory and degenerative tissue pathologies and represents an effective tool in the treatment of early and intermediate osteoarthritis. To date, the demonstration of the efficacy of BB-02 therapy has been measured through the evaluation of clinical endpoints, using both objective and subjective assessment scales. So far, there is a lack of instrumental measurement of the ability of BB-02 therapy to preserve the integrity of the articular cartilage.

The primary objective of the study is to evaluate, through magnetic resonance imaging (MRI), the effect of pulsed electromagnetic fields administered via BB-02 therapy on cartilage damage in subjects with early-stage osteoarthritis. The BB-02 device was chosen based on promising results reported in the pre-clinical phase of experimentation.

The secondary objective is to assess the effect of BB-02 therapy on pain resolution and clinical scores of knee functionality in the two different therapeutic regimens.

DETAILED DESCRIPTION:
Knee osteoarthritis (gonarthrosis) is an extremely debilitating condition for affected patients, who experience progressive functional limitations with consequent impairment of daily activities and quality of life. Additionally, this condition represents a significant burden on the national healthcare system due to the severe functional limitations of affected patients and the high costs of interventions and devices used for prosthetic replacement. Knee replacement surgery is the gold standard treatment for gonarthrosis; however, this procedure carries a doubled risk of failure in patients under 60 years of age. Therefore, considering the high number of patients affected by early or intermediate-stage osteoarthritis at an age characterized by high functional demands, it becomes essential to identify treatment alternatives aimed primarily at resolving symptoms but also at slowing down the degenerative joint process, with the goal of delaying the need for prosthetic treatment as much as possible.

While various surgical solutions, including joint preservation procedures, have been proposed, clear evidence is still lacking regarding the effectiveness of conservative treatments in protecting and possibly regenerating the pathological articular cartilage that characterizes patients with gonarthrosis. In this scenario, quantifying the therapeutic potential of non-surgical treatment devices for patients with gonarthrosis is of considerable importance in the development of degenerative joint disease treatment. From this need arises the desire to verify the regenerative potential of available strategies for the treatment of joint pathologies.

Biophysical stimulation with variable intensity magnetic fields over time represents a therapeutic option supported by a solid body of scientific literature for the treatment of conditions associated with joint osteoarthritis such as bone edema and soft tissue distress. The medical device BB-02 (IGEA SpA, Carpi, Italy) is a certified medical device according to Regulation (EU) 2017/745 (MDR) for the treatment of inflammatory and degenerative tissue diseases. BB-02 is used for inflammation control and chondroprotection: chondroprotection refers to the set of pharmacological, physical, surgical, alone or combined treatments, aimed at preserving cartilage integrity or limiting damage due to degenerative, pathological, and traumatic processes, as well as inflammatory reactions. BB-02 therapy limits the degenerative effects of inflammation present in the joint environment after trauma or surgery. The medical device BB-02 extinguishes joint inflammation through an adenosine agonist action on the A2A receptor and exerts a strong chondroprotective effect. Extensive translational research has shown that biophysical stimulation with BB-02 therapy is capable of modulating cartilage metabolism (Massari L 2007).

In vitro, BB-02 therapy induces a significant increase in both chondrocyte proliferation in the presence of growth factors, such as IGF-1, and proteoglycan synthesis, even in the presence of inflammatory phenomena, such as IL-1β (De Mattei M 2003, 2004, 2009; Ongaro A 2011, Veronesi 2015). In vitro studies on neutrophils, synoviocytes, and chondrocytes have shown that BB-02 therapy increases the availability of adenosine A2A receptors and, acting as chondroprotective agents, reduces tissue damage due to the inflammatory response (Varani K, 2002, 2008, 2017). Stimulation with BB-02 therapy, by reducing the release of inflammation mediators involved in cartilage degeneration, such as inflammatory cytokines (IL-6 and IL-8) and lipid mediators of inflammation (prostaglandin E2), enhances the anti-inflammatory effect of individual adenosinic agonists A2A and A3 by increasing the release of anti-inflammatory cytokines such as IL-10 (Ongaro A 2012, Vincenzi F 2013). Synovial stem cells have shown a high chondrogenic potential; in culture, with appropriate chondroinductive supplements supplemented with TGF-β3, they are capable of differentiating in a chondrogenic direction. In a study conducted on these types of cells, chondrogenic differentiation was analyzed in the presence of inflammatory conditions, obtained by adding the culture medium with IL-1β (Ongaro A 2015), and BB-02 therapy. Stimulation is able to inhibit the inflammatory phenomenon and preserve the chondrocyte phenotype. These and other results have been confirmed in animal models of osteoarthritis where stimulation with BB-02 therapy has led to a reduction in the progression of osteoarthritic lesions in the knee (Fini M 2005, 2008, Veronesi F 2014). In sheep undergoing osteochondral transplantation, BB-02 therapy was able to promote the formation of new subchondral bone tissue, reducing areas of bone resorption, avoiding complete implant resorption (Benazzo F 2008). Evidence of an anabolic and trophic effect has been observed with high synthesis of anabolic factors, such as TGF-β, and inhibition of the synthesis of pro-inflammatory cytokines, such as TNF-α and IL-1β. In rabbits with osteochondral lesions, BB-02 therapy has been shown to be effective in significantly improving the quality of regenerated tissue, both bone and cartilage, in osteochondral defects in the presence of collagen scaffolds and bone marrow concentrate (BMC) (Veronesi F BMC Musculoskelet Disord. 2015). The anti-inflammatory activity of BB-02 therapy effectively counteracts the degenerative effect of IL-1β, significantly improving cartilage regeneration compared to non-stimulated lesions. Recently, the Columbia University group has demonstrated how BB-02 therapy is able to maximize the survival and functionality of osteochondral implants in tissue engineering methods (Stefani RM 2020). In clinical practice, in the conservative treatment of joint pathologies such as Bone Marrow Edema (Martinelli N 2015, Perugia D 2015), spontaneous osteonecrosis of the knee (Marcheggiani Muccioli G 2012), early-stage knee osteoarthritis (Gobbi A 2013), and patellofemoral pathology (Immarrone CS 2016), BB-02 therapy has been shown to be effective in resolving the area of bone marrow edema and improving joint functional recovery. Imaging diagnostics in the study of cartilage pathology can non-invasively confirm the presence of cartilage pathology, establish the degree of alterations, enable proper therapy planning (conservative or surgical), and verify its effectiveness over time. Conventional radiography (X-ray) is the most basic and cost-effective imaging technique and is used as a first-level investigation in the diagnosis of degenerative joint pathology, but it is of limited use in evaluating early stages and initial alterations of articular cartilage. The advent of magnetic resonance imaging (MRI), with its superior soft tissue contrast and multiplanar imaging capabilities, has solved many problems in imaging articular cartilage, providing non-invasive, both morphological and biochemical, information on the cartilage state. Morphological information provided by MRI includes both focal and diffuse cartilage lesions. MRI provides information such as thickness, volume, and three-dimensional morphology of the cartilage; biochemical information is represented by the ability to determine the content of water, proteoglycans, and collagen. Knowledge of this additional information is of great utility in understanding cartilage pathology and therefore in choosing therapeutic treatment.

In this study, we aim to evaluate the efficacy of two different therapeutic regimens with BB-02 therapy in patients still active in sports with initial cartilage damage. The present study aims to observe the effect of BB-02 therapy on cartilage through high-field MRI (3 Tesla, 3T) investigation capable of providing both morphological and biochemical information on joint structures. With 3T MRI, we will evaluate the knee articular cartilage before and after treatment, focusing on initial superficial lesions present before treatment, and at the end of therapy, assessing whether and to what extent they are repaired.

Two different therapeutic regimens of BB-02 therapy will be applied in the study: 4 hours a day for 30 days and 1 hour a day for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes aged between 20 and 55 years.
* Body Mass Index, BMI < 35.
* Subjects with Kellgren-Lawrence grade 2 osteoarthritis.
* Subjects with baseline Visual Analog Scale (VAS) score ≥ 2.
* Mechanical alignment between 175° and 185°.
* Absence of acute ligamentous or meniscal pathology.

Exclusion Criteria:

* Patients with systemic inflammatory or neoplastic diseases
* Smokers
* Individuals with hypertension or diabetes
* Knee arthroscopy within the 12 months prior to enrollment
* Subjects diagnosed with inflammatory arthritis (rheumatoid arthritis, gout, joint infections, Lyme disease, lupus, etc.)
* Subjects diagnosed with secondary arthritis (acromegaly, Charcot arthropathy, hemochromatosis, Wilson's disease, ochronosis, anterior cruciate ligament injuries)
* Patients undergoing analgesic therapy with opioids, systemic corticosteroids, or intra-articular corticosteroids during study participation
* Patients undergoing intra-articular injections of hyaluronic acid during the study participation
* Patients unable to provide informed consent
* Pregnant and breastfeeding women
* Women in menopause

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
3 Tesla Magnetic Resonance Imaging (MRI) | 12 months
  with T2 mapping sequences in patients with knee osteoarthritis before and after treatment with two different therapeutic regimens of BB-02 therapy

SECONDARY OUTCOMES:
visual analog scale (vas) | 12 months
  It is a one-dimensional quantitative numeric pain rating scale with 10 points; the scale requires the patient to select the number that best describes the intensity of their pain, from 0 to 10, at the time of the visit and before the surgery. 0 means no pain and 10 indicates the worst possible pain.
Knee Society Score (KSS) | 12 months
  The Knee Society Score (KSS) is a comprehensive system used to evaluate knee joint condition and functionality, especially before and after knee replacement surgery. It consists of two parts: the Knee Score, assessing pain, range of motion, stability, and alignment, and the Function Score, evaluating the patient's ability to perform daily activities like walking and climbing stairs. Both scores can reach up to 100 points, with higher scores indicating better knee health and function. KSS is widely used to assess surgical outcomes and track patient progress.
Tegner Activity Score (TAS) | 12 months
  It allows for estimating the level of motor activity of an individual with a score between 0 and 10, where 0 represents ''incapacity'' and 10 represents ''participation in competitive sports, such as national or international level soccer.' This score is the most commonly used to define the level of motor activity in patients with knee disorders. The patient will also be asked how many years they have been active in sports and whether the cause of reduction or cessation of activity is related to their knee condition or not.
Degree of patient compliance with the treatment | 12 months
  The patient's ability to adhere correctly, in methods and timing, to a therapy indicated by their doctor, without the possibility of altering the therapeutic treatment in order to comply with the study group and the clinical protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Result] Adravanti P, Nicoletti S, Setti S, Ampollini A, de Girolamo L. Effect of pulsed electromagnetic field therapy in patients undergoing total knee arthroplasty: a randomised controlled trial. Int Orthop. 2014 Feb;38(2):397-403. doi: 10.1007/s00264-013-2216-7. Epub 2013 Dec 20. PMID 24352823
- [Result] Benazzo F, Cadossi M, Cavani F, Fini M, Giavaresi G, Setti S, Cadossi R, Giardino R. Cartilage repair with osteochondral autografts in sheep: effect of biophysical stimulation with pulsed electromagnetic fields. J Orthop Res. 2008 May;26(5):631-42. doi: 10.1002/jor.20530. PMID 18176941
- [Result] Cadossi M, Buda RE, Ramponi L, Sambri A, Natali S, Giannini S. Bone marrow-derived cells and biophysical stimulation for talar osteochondral lesions: a randomized controlled study. Foot Ankle Int. 2014 Oct;35(10):981-7. doi: 10.1177/1071100714539660. Epub 2014 Jun 10. PMID 24917648
- [Result] Moretti L, Bizzoca D, Giancaspro GA, Cassano GD, Moretti F, Setti S, Moretti B. Biophysical Stimulation in Athletes' Joint Degeneration: A Narrative Review. Medicina (Kaunas). 2021 Nov 4;57(11):1206. doi: 10.3390/medicina57111206. PMID 34833424
- [Result] Perdisa F, Bordini B, Salerno M, Traina F, Zaffagnini S, Filardo G. Total Knee Arthroplasty (TKA): When Do the Risks of TKA Overcome the Benefits? Double Risk of Failure in Patients up to 65 Years Old. Cartilage. 2023 Sep;14(3):305-311. doi: 10.1177/19476035231164733. Epub 2023 Apr 19. PMID 37073516